CLINICAL TRIAL: NCT04864249
Title: The Impact of a Neonatal Sleep Intervention on Postpartum Blood Pressure in Women With Hypertensive Disorders of Pregnancy
Brief Title: Neonatal Sleep Intervention to Improve Postpartum Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alisse Hauspurg (Other)
Collaborators: Happiest Baby, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Alisse Hauspurg, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20070054
Record Dates: First submitted 2021-04-24; First posted 2021-04-28 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Pre-Eclampsia; Gestational Hypertension; Sleep
Keywords: Pre-Eclampsia; Gestational Hypertension; Postpartum Sleep; SNOO
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SNOO Responsive Bassinet (Experimental): Will receive and be instructed on the use of the SNOO responsive bassinet for their newborn + the current standard of care of safe sleep education in the postpartum period
  Interventions: Device: SNOO; Other: Safe sleep education in the postpartum period
- Usual Care (Active Comparator): Will receive the current standard of care of safe sleep education in the postpartum period
  Interventions: Other: Safe sleep education in the postpartum period

INTERVENTIONS:
Device: SNOO — The SNOO is a commercially available device which is a responsive bassinet for neonates. The bassinet is designed to respond to the infant's cries and automatically respond by emitting engineered white noise sounds and providing a rhythmic rocking motion. The infant is also swaddled to remain securely back-down. The SNOO automatically increases the emitted sound and motion if the infant is still crying. However, if the infant does not settle within 3 minutes, the SNOO will shut off and alert the adults for additional assistance. Parents can also modify the SNOO settings to meet the baby's need for sound and/or motion.
  Arms: SNOO Responsive Bassinet
Other: Safe sleep education in the postpartum period — Comprised of education from the postpartum clinical nurse with a corresponding educational handout to take home

SUMMARY:
The investigators are conducting a single center, randomized controlled trial testing the impact of a neonatal sleep intervention, the SNOO, on reducing maternal blood pressure (BP) in the postpartum period in women with hypertensive disorders of pregnancy. The SNOO is a responsive bassinet designed to automatically calm and consolidate infants by responding to their cries. Use of the SNOO has been demonstrated to improve infant sleep by 1-2 hours nightly, thus increasing maternal sleep time. The investigators plan for 110 women with pregnancies complicated by gestational hypertension or pre-eclampsia to be randomized 1:1 to either receive and use the SNOO responsive bassinet for their infants, or to receive the usual care of safe sleep education. Women will be followed longitudinally through 6 months postpartum with serial BPs, weights, mood assessments, and subjective and objective sleep assessments. The investigators hypothesize that for women with pregnancies complicated by gestational hypertension or preeclampsia, that poor maternal sleep quality contributes to increased BP in the postpartum period. The investigators further propose that compared to usual care (safe sleep education), an intervention targeted to improve neonatal sleep (the SNOO), and thus maternal sleep, will improve postpartum BP for these women.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Have a singleton, full-term (37 or greater weeks of gestation), live birth of a non-anomalous fetus
* Diagnosis of gestational hypertension or pre-eclampsia by American College of Obstetricians and Gynecologists criteria
* Enrolled in the institution's postpartum blood pressure remote monitoring program
* Willing to undergo randomization
* Willing to use the SNOO for their neonate in the postpartum period if randomized to that study arm

Exclusion Criteria:

* <18 years old
* Non-English speaking
* Diagnosis of chronic hypertension
* Diagnosis of pre-gestational diabetes
* Diagnosis of cardiac disease
* Diagnosis of kidney disease
* Diagnosis of liver disease
* Infant admitted to the neonatal intensive care unit
* Intend to use the SNOO prior to study enrollment
* Not willing to be randomized
* Not willing to use the SNOO if randomized to that study arm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alisse Hauspurg, MD, Principal Investigator — University of Pittsburgh, Magee-Womens Hospital
Locations (1):
- University of Pittsburgh Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang TL, Quinn BA, Hart R, Wiener AA, Facco FL, Simhan HN, Hauspurg AK. The effect of a neonatal sleep intervention on maternal postpartum hypertension: a randomized trial. Am J Obstet Gynecol MFM. 2024 Feb;6(2):101239. doi: 10.1016/j.ajogmf.2023.101239. Epub 2023 Dec 10. PMID 38072236

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SNOO Responsive Bassinet | Usual Care
Started | 54 | 56
Completed | 45 | 31
Not Completed | 9 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SNOO Responsive Bassinet | Usual Care | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (5.5) | 30.5 (4.8) | 31.1 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 56 | 110
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 53 | 54 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Self-reported race: Black | 10 | 10 | 20
  Self-reported race: White | 43 | 41 | 84
  Self-reported race: Asian or Pacific Islander | 1 | 2 | 3
  Self-reported race: Other | 0 | 3 | 3
Partner status [Count of Participants; unit: Participants]
  Married or partnered | 49 | 43 | 92
  Separated or divorced | 0 | 2 | 2
  Single | 5 | 11 | 16
Annual household income [Count of Participants; unit: Participants]
  <$75,000 | 21 | 26 | 47
  $75,000+ | 31 | 24 | 55
  Prefer not to answer | 2 | 6 | 8
Insurance status during pregnancy [Count of Participants; unit: Participants]
  Private | 42 | 36 | 78
  Public | 9 | 17 | 26
  Other | 1 | 1 | 2
  No insurance | 2 | 2 | 4
Other children also living at home [Count of Participants; unit: Participants] | 25 | 23 | 48
Smoking within the past 2 years [Count of Participants; unit: Participants] | 6 | 8 | 14
Pre-delivery diagnosis of depression [Count of Participants; unit: Participants] | 17 | 18 | 35
Ever breastfeed [Count of Participants; unit: Participants] | 48 | 49 | 97
Gestational age at delivery [Median (Inter-Quartile Range); unit: weeks] | 38.1 [37.3 to 39.0] | 38.1 [37.4 to 39.2] | 38.1 [37.4 to 39.1]
Mode of delivery [Count of Participants; unit: Participants]
  Vaginal delivery | 35 | 31 | 66
  Forceps-assisted vaginal delivery | 1 | 1 | 2
  Vacuum-assisted vaginal delivery | 0 | 3 | 3
  Cesarean delivery | 18 | 21 | 39
Blood loss during delivery [Median (Inter-Quartile Range); unit: mL] | 300 [200 to 550] | 300 [150 to 500] | 300 [200 to 500]
Neonatal birthweight [Median (Inter-Quartile Range); unit: g] | 3155 [2915 to 3700] | 3055 [2685 to 3305] | 3125 [2830 to 3430]
Type of hypertensive disorder [Count of Participants; unit: Participants] — The diagnoses of gestational hypertension, preeclampsia without severe features, and preeclampsia with severe features were based on criteria established by the American College of Obstetricians and Gynecologists (ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1.)
  Participants
    Gestational hypertension | 24 | 33 | 57
    Preeclampsia without severe features | 15 | 11 | 26
    Preeclampsia with severe features | 15 | 12 | 27
Gestational age at diagnosis of hypertensive disorder [Median (Inter-Quartile Range); unit: weeks] | 38.0 [36.4 to 38.7] | 37.9 [36.4 to 39.1] | 37.9 [36.4 to 39]
Mean arterial pressure at first prenatal visit [Mean (Standard Deviation); unit: mm Hg] — The mean arterial pressure at the first prenatal visit represents a baseline measure assessing one component of the participant's health early in pregnancy prior to the onset of any hypertensive disorder of pregnancy. Population: Some participant data not available in chart review
  mm Hg
    number analyzed (Participants) | 54 | 54 | 108
    (all) | 87 (7) | 90 (8) | 89 (8)
Systolic blood pressure at first prenatal visit [Mean (Standard Deviation); unit: mm Hg] — The systolic blood pressure at the first prenatal visit represents a baseline measure assessing one component of the participant's health early in pregnancy prior to the onset of any hypertensive disorder of pregnancy. Population: Some participant data not available in chart review
  mm Hg
    number analyzed (Participants) | 54 | 54 | 108
    (all) | 115 (10) | 119 (9) | 118 (10)
Diastolic blood pressure at first prenatal visit [Mean (Standard Deviation); unit: mm Hg] — The diastolic blood pressure at the first prenatal visit represents a baseline measure assessing one component of the participant's health early in pregnancy prior to the onset of any hypertensive disorder of pregnancy. Population: Some participant data not available in chart review
  mm Hg
    number analyzed (Participants) | 54 | 54 | 108
    (all) | 73 (8) | 76 (9) | 74 (9)
Weight in kg at first prenatal visit [Median (Inter-Quartile Range); unit: kg] — The weight at the first prenatal visit represents a baseline measure assessing one component of the participant's health early in pregnancy prior to the onset of any hypertensive disorder of pregnancy. Population: Some participant data not available in chart review
  kg
    number analyzed (Participants) | 54 | 54 | 108
    (all) | 74.8 [65.3 to 90.7] | 81.0 [66.5 to 96.5] | 76.3 [65.6 to 94.8]
Body Mass Index in kg/m^2 at first prenatal visit [Median (Inter-Quartile Range); unit: kg/m^2] — The Body Mass Index at the first prenatal visit represents a baseline measure assessing one component of the participant's health early in pregnancy prior to the onset of any hypertensive disorder of pregnancy. Population: Some participant data not available in chart review
  kg/m^2
    number analyzed (Participants) | 54 | 54 | 108
    (all) | 27.7 [24.0 to 35.8] | 30.0 [25.2 to 35.2] | 29.1 [25.0 to 35.4]
Mean arterial pressure on Labor and Delivery admission [Mean (Standard Deviation); unit: mm Hg] | 103 (12) | 102 (9) | 103 (11)
Systolic blood pressure on Labor and Delivery admission [Mean (Standard Deviation); unit: mm Hg] | 140 (13) | 135 (12) | 138 (13)
Diastolic blood pressure on Labor and Delivery admission [Mean (Standard Deviation); unit: mm Hg] | 86 (13) | 86 (10) | 86 (12)
Weight on Labor and Delivery admission in kg [Median (Inter-Quartile Range); unit: kg] | 90.9 [79.0 to 104.0] | 93.5 [78.3 to 111.5] | 91.6 [78.5 to 108.2]
Body Mass Index on Labor and Delivery admission in kg/m^2 [Median (Inter-Quartile Range); unit: kg/m^2] | 33.8 [29.5 to 39.3] | 35.5 [30.2 to 40.6] | 34.9 [29.9 to 40.4]
Mean arterial pressure at postpartum enrollment [Mean (Standard Deviation); unit: mm Hg] | 102 (8) | 102 (11) | 102 (10)
Systolic blood pressure at postpartum enrollment [Mean (Standard Deviation); unit: mm Hg] | 135 (12) | 134 (14) | 135 (13)
Diastolic blood pressure at postpartum enrollment [Mean (Standard Deviation); unit: mm Hg] | 85 (8) | 86 (10) | 86 (9)
Number of participants on antihypertensive medication(s) at postpartum enrollment [Count of Participants; unit: Participants] — Whether or not the participant is taking antihypertensive medication(s) for blood pressure control will be assessed at the time of postpartum enrollment.
  Participants | 4 | 3 | 7
Number of participants with Stage 1+ hypertension or on antihypertensive medication(s) [Count of Participants; unit: Participants] — Whether or not the participant meets criteria for Stage 1 or greater hypertension or is taking antihypertensive medication(s) for blood pressure control will be assessed at the time of postpartum enrollment. The American College of Cardiology categorizes blood pressure into normal, elevated, Stage 1, Stage 2, or hypertensive crisis, with hypertensive crisis being the most severe. Stage 1 hypertension was defined as a systolic blood pressure of ≥130 and/or or diastolic blood pressure of ≥80.
  Participants | 9 | 11 | 20
Weight at postpartum enrollment in kg [Median (Inter-Quartile Range); unit: kg] | 87.2 [74.8 to 103.4] | 92.7 [75.6 to 107.5] | 88.6 [75.2 to 106.8]
Body Mass Index at postpartum enrollment in kg/m^2 [Median (Inter-Quartile Range); unit: kg/m^2] | 32.2 [27.7 to 39.5] | 34.5 [28.5 to 39.7] | 33.2 [28.2 to 39.5]

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Pressure
Description: Mean arterial pressure will be calculated from the systolic and diastolic blood pressures [(2 * diastolic blood pressure + systolic blood pressure) / 3] assessed using a study-provided blood pressure cuff at the time of the study follow-up visit.
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 51
mm Hg | 93 (8) | 94 (8)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.54, t-test, 2 sided

2. Secondary Outcome: Mean Arterial Pressure
Description: as for outcome 1
Time Frame: 1 week postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 49
mm Hg | 99 (10) | 103 (7)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.04, t-test, 2 sided

3. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure will be assessed using a study-provided blood pressure cuff at the time of the study follow-up visit
Time Frame: 1 week postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 49
mm Hg | 131 (14) | 130 (10)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.89, t-test, 2 sided

4. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure will be assessed using a study-provided blood pressure cuff at the time of the study follow-up visit
Time Frame: 1 week postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 49
mm Hg | 83 (11) | 89 (8)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.003, t-test, 2 sided

5. Secondary Outcome: Number of Participants on Antihypertensive Medication(s)
Description: Whether or not the participant is taking antihypertensive medication(s) for blood pressure control will be assessed at the time of the study follow-up visit.
Time Frame: 1 week postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 49
Participants | 12 | 19
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.15, Chi-squared

6. Secondary Outcome: Number of Participants With Stage 1+ Hypertension or on Antihypertensive Medication(s)
Description: Whether or not the participant meets criteria for Stage 1 or greater hypertension or is taking antihypertensive medication(s) for blood pressure control will be assessed at the time of the study follow-up visit. The American College of Cardiology categorizes blood pressure into normal, elevated, Stage 1, Stage 2, or hypertensive crisis, with hypertensive crisis being the most severe. Stage 1 hypertension was defined as a systolic blood pressure of ≥130 and/or or diastolic blood pressure of ≥80.
Time Frame: 1 week postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 49
Participants | 43 | 44
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.84, Chi-squared

7. Secondary Outcome: Maternal Weight in Kilograms
Description: Maternal weight in kilograms will be assessed using a study-provided scale at the time of the study follow-up visit
Time Frame: 1 week postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 49
kg | 81.2 [70.6 to 94.3] | 88.0 [69.8 to 104.1]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Body Mass Index in kg/m^2
Description: Body mass index in kg/m^2 will be assessed at the time of the study follow-up visit
Time Frame: 1 week postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 49
kg/m^2 | 29.4 [26.3 to 39.8] | 31.6 [28.0 to 37.9]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.55, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Systolic Blood Pressure
Description: as for outcome 3
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 51
mm Hg | 121 (10) | 122 (11)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.55, t-test, 2 sided

10. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 4
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 51
mm Hg | 79 (8) | 80 (8)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.62, t-test, 2 sided

11. Secondary Outcome: Number of Participants on Antihypertensive Medication(s)
Description: as for outcome 5
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 51
Participants | 8 | 13
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.19, Chi-squared

12. Secondary Outcome: Number of Participants With Stage 1+ Hypertension or on Antihypertensive Medication(s)
Description: as for outcome 6
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 51
Participants | 31 | 32
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.66, Chi-squared

13. Secondary Outcome: Maternal Weight in Kilograms
Description: Maternal weight in kilograms will be assessed using a study-provided scale at the time of the study follow-up visit
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 51
kg | 76.7 [69.0 to 93.6] | 87.0 [69.4 to 103.4]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Body Mass Index
Description: Body mass index in kg/m^2 will be assessed at the time of the study follow-up visit
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 53 | 51
kg/m^2 | 28.5 [25.7 to 35.4] | 32.1 [26.2 to 37.6]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Mean Arterial Pressure
Description: as for outcome 1
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 45 | 31
mm Hg | 93 (9) | 94 (8)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.56, t-test, 2 sided

16. Secondary Outcome: Systolic Blood Pressure
Description: as for outcome 3
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 45 | 31
mm Hg | 121 (10) | 122 (12)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.80, t-test, 2 sided

17. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 4
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 45 | 31
mm Hg | 78 (10) | 80 (7)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.48, t-test, 2 sided

18. Secondary Outcome: Number of Participants on Antihypertensive Medication(s)
Description: as for outcome 5
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 45 | 31
Participants | 3 | 3
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.62, Chi-squared

19. Secondary Outcome: Number of Participants With Stage 1+ Hypertension or on Antihypertensive Medication(s)
Description: as for outcome 6
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 45 | 31
Participants | 21 | 19
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.21, Chi-squared

20. Secondary Outcome: Maternal Weight in Kilograms
Description: Maternal weight in kilograms will be assessed using a study-provided scale at the time of the study follow-up visit
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 45 | 31
kg | 77.2 [67.1 to 87.1] | 85.8 [68.5 to 102.1]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Body Mass Index in kg/m^2
Description: Body mass index in kg/m^2 will be assessed at the time of the study follow-up visit
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 45 | 31
kg/m^2 | 27.8 [25.0 to 34.7] | 31.6 [25.8 to 36.5]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Pittsburgh Sleep Quality Index Score
Description: The Pittsburgh Sleep Quality Index contains 19 self-rated questions and 5 questions rated by the bed partner or roommate if one is available; only the self-rated questions are included in the scoring. Scores range from 0 (indicating no difficulties in any aspect of sleep) to 21 (indicating severe difficulties in all areas).
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 48 | 34
score on a scale | 8.5 (3.0) | 8.9 (3.2)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.51, t-test, 2 sided

23. Secondary Outcome: PROMIS Sleep Disturbance Questionnaire
Description: The PROMIS Sleep Disturbance Questionnaire contains 27 self-rated questions on subjective sleep quality. Scores range from 27 (indicating excellent sleep quality) to 135 (indicating poor sleep quality).
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 48 | 34
units on a scale | 55 (17) | 58 (19)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.38, t-test, 2 sided

24. Secondary Outcome: Epworth Sleepiness Scale Score
Description: The Epworth Sleepiness Scale contains 8 self-rated questions to determine the level of daytime sleepiness in individuals. Scores range from 0 to 24. A score of 10 or more is concerning for excessive daytime sleepiness.
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 48 | 34
score on a scale | 8.3 (4.1) | 7.9 (3.7)
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.68, t-test, 2 sided

25. Secondary Outcome: Edinburgh Postnatal Depression Scale Score
Description: The Edinburgh Postnatal Depression Scale contains 10 self-rated questions to assess for major depression in the postnatal period. Scores range from 0 to 30. A score of 13 or greater is concerning for major depression.
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 48 | 34
score on a scale | 5 [2 to 9] | 3 [1 to 8]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.42, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Generalized Anxiety Disorder 2-item Score
Description: The Generalized Anxiety Disorder 2-item contains 2 self-rated questions to screen for generalized anxiety disorder. Scores range from 0 to 6. A score of 3 or greater is concerning for generalized anxiety disorder.
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 48 | 34
score on a scale | 1 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Perceived Stress Scale 4 Score
Description: The Perceived Stress Scale 4 contains 4 self-rated questions regarding stress levels. Scores range from 0 to 16. Higher scores a correlated to more stress.
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 48 | 34
score on a scale | 3.5 [2 to 5] | 3.5 [2 to 5.5]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Breslau 7-Item Screen for Post-traumatic Stress Disorder Score
Description: The Breslau 7-Item Screen for Posttraumatic Stress Disorder contains 7 self-rated questions assessing symptoms of post-traumatic stress disorder. Scores range from 0 to 7. Scores of 4 or above are concerning for post-traumatic stress disorder.
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 48 | 34
score on a scale | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: Median Infant Total Daily Sleep
Description: Participants will be asked to self-complete 7 days of an infant sleep log in the 7 days prior to the study follow-up visit. The median total daily sleep in hours per day will be calculated over the 7 days of sleep log data recorded.
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: hours per day
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 42 | 22
hours per day | 13.6 [12.1 to 14.9] | 13.7 [13.0 to 15.0]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Median Infant Daily Longest Sleep Duration
Description: Participants will be asked to self-complete 7 days of an infant sleep log in the 7 days prior to the study follow-up visit. The median daily longest sleep duration in hours per day will be calculated over the 7 days of sleep log data recorded.
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: hours per day
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 42 | 22
hours per day | 4.0 [3.5 to 4.6] | 4.0 [3.1 to 4.4]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: Median Maternal Total Daily Sleep
Description: Participants will be asked to self-complete 7 days of a maternal sleep log in the 7 days prior to the study follow-up visit. The median total daily sleep in hours per day will be calculated over the 7 days of sleep log data recorded.
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: hours per day
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 42 | 22
hours per day | 6.4 [5.9 to 7.7] | 7.4 [6.9 to 7.9]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: Median Maternal Daily Longest Sleep Duration
Description: Participants will be asked to self-complete 7 days of a maternal sleep log in the 7 days prior to the study follow-up visit. The median daily longest sleep duration in hours per day will be calculated over the 7 days of sleep log data recorded.
Time Frame: 6 weeks postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: hours per day
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 42 | 22
hours per day | 3.4 [2.8 to 4.1] | 3.6 [3.1 to 4.9]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney)

33. Secondary Outcome: Median Infant Total Daily Sleep
Description: as for outcome 29
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: hours per day
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 41 | 20
hours per day | 13.2 [11.9 to 13.9] | 13.5 [12.8 to 14.1]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney)

34. Secondary Outcome: Median Infant Daily Longest Sleep Duration
Description: as for outcome 30
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: hours per day
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 41 | 20
hours per day | 7.7 [5.6 to 8.9] | 6.5 [5.2 to 7.7]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: Median Maternal Total Daily Sleep
Description: as for outcome 31
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: hours per day
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 41 | 20
hours per day | 7.3 [6.2 to 8.0] | 7.8 [6.9 to 8.2]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Median Maternal Daily Longest Sleep Duration
Description: as for outcome 32
Time Frame: 4 months postpartum
Population: Some participants lost to follow-up and/or did not complete this outcome measure
Measure: Median (Inter-Quartile Range); unit: hours per day
Arm/Group | SNOO Responsive Bassinet | Usual Care
Number analyzed (Participants) | 41 | 20
hours per day | 5.9 [4.3 to 7.1] | 5.1 [4.2 to 6.9]
Statistical Analysis 1: Comparison: SNOO Responsive Bassinet vs Usual Care; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SNOO Responsive Bassinet | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/56
Other Adverse Events (participants affected / at risk) | 0/54 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT04864249/Prot_SAP_000.pdf